CLINICAL TRIAL: NCT03774836
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Three-Arm Study to Evaluate the Efficacy and Safety of Tramadol Infusion (AVE-901) Versus Placebo and Morphine in the Management of Postoperative Pain Following Abdominoplasty
Brief Title: Tramadol Versus Placebo and Morphine in the Management of Post-Operative Pain Abdominoplasty
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Avenue Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AVE-901-103
Record Dates: First submitted 2018-12-11; First posted 2018-12-13 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-02

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia | interventions — Tramadol; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Tramadol 50 mg (Active Comparator): Given at Hours 0, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, and 44
  Interventions: Drug: Tramadol
- Morphine 4 mg (Active Comparator): Given at Hours 0, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, and 44
  Interventions: Drug: Morphine
- Placebo (Placebo Comparator): Given at Hours 0, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, and 44
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tramadol — IV Tramadol 50 mg, given at Hours 0, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, and 44
  Arms: Tramadol 50 mg
Drug: Morphine — Morphine 4 mg, given at Hours 0, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, and 44
  Arms: Morphine 4 mg
Other: Placebo — Placebo, given at Hours 0, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, and 44
  Arms: Placebo

SUMMARY:
This study is evaluating the analgesic efficacy of intravenous (IV) tramadol (AVE-901) compared to placebo in the management of postoperative pain following abdominal surgery.

DETAILED DESCRIPTION:
(Non-clinical summary) Tramadol is a centrally-acting synthetic analgesic of the aminocyclohexanol group with opioid-like effects. Tramadol is extensively metabolized following administration, which results in a number of enantiomeric metabolites that display different opioid-receptor binding properties, and monoaminergic reuptake inhibition.

ELIGIBILITY:
Inclusion Criteria:

* The patient is male or female 18-75 years of age
* Willing to give consent and able to understand the study procedures
* Female patients must be of non-childbearing potential or be practicing a highly effective contraption
* The patient must be willing to be housed in a healthcare facility and able to receive parenteral analgesia for at least 48 hours after surgery
* The patient meets definition of American Society of Anesthesiologists (ASA) Physical Class 1, or 2.

Exclusion Criteria:

* The patient is undergoing an abdominoplasty of significant complexity defined as pre-planned surgical time of greater than 180 mins.
* The patient has a recent (within 5 years) and/or current history of chronic analgesic, opiate or tranquilizer abuse or dependence or is a user of illicit drugs or has had a recent history (within 2 years) of drug or alcohol abuse.
* The patient is taking herbal or dietary supplements or medications that are moderate or strong inhibitors of CYP2D6 or CYP3A4 (e.g., fluoxetine, paroxetine, amitriptyline, quinidine, ketoconazole, erythromycin, grapefruit juice) or inducers of CYP3A4 (e.g., carbamazepine, rifampin, St. John's Wort) and cannot go through a minimum washout period of 14 days prior to surgery.
* The patient has a history of epilepsy, is susceptible to seizures.
* The patient cannot be withdrawn from medications (at least 7 days prior to surgery) that may lower the seizure threshold (e.g. anti-psychotic agents, MAOI inhibitors) or which increase serotonergic tone (e.g. selective serotonin reuptake inhibitors (SSRIs), serotonin norepinephrine reuptake inhibitors (SNRIs), tricyclic antidepressants, triptans, cyclobenzaprine triptans).
* The patient has had a recent cardiovascular event or clinically significant abnormal ECG finding at screening or baseline.
* The patient has a history of Long QT Syndrome or a relative with this condition.
* The patient has expressed suicidal ideation or is considered to be at risk of suicide.
* The patient is morbidly obese (body mass index [BMI] ≥ 40 kg/m2) or has documented sleep apnea requiring CPAP or other treatment.
* Female patient is pregnant and/or undergoing a pregnancy-related surgery, or breastfeeding.
* The patient has a history of cardiopulmonary, neurological or psychiatric or other medical condition that may confound the assessments of efficacy or safety.
* The patient has cirrhosis, moderate or severe hepatic impairment or an alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value > 3X upper limit of normal (ULN) at Screening.
* The patient has severe renal impairment or a serum creatinine value of > 2.0 mg/dL at Screening.
* The patient has potassium, sodium, calcium or magnesium levels outside of the normal range or any other clinically significant abnormalities in laboratory values at Screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2018-12-14 (Actual); Primary Completion 2019-05-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
The Sum of Pain Intensity Differences through 24 hours | 24 hours post dose

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Lotus Clinical Research, Pasadena, California
  - Hermann Drive Research, Houston, Texas
  - Endeavor Clinical Trials, San Antonio, Texas